CLINICAL TRIAL: NCT00034359
Title: A Double-Blind, Randomized Trial of Antiviral Activity and Safety of 12 Weeks Oral Treatment With ACH-126,443 (Beta-L-Fd4C) in Treatment-Naive HBV-Infected Adults
Brief Title: Safety and Antiviral Activity Study of ACH-126,443 (Beta-L-Fd4C) in Treatment-naive Adults With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACH443-003
Record Dates: First submitted 2002-04-26; First posted 2002-04-29 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Hepatitis B, Chronic
Keywords: E-antigen Positive; Treatment-naive Chronic Hepatitis B; Achillion
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — dexelvucitabine; Lamivudine

INTERVENTIONS:
Drug: ACH-126,443
  Other Names: beta-L-Fd4C
Drug: Lamivudine
Drug: Placebo

SUMMARY:
The purpose of this study was to determine the safety and anti-hepatitis B virus (-HBV) activity of ACH-126,443 in comparison to lamivudine or placebo in treatment-naive adults with chronic hepatitis B infection.

DETAILED DESCRIPTION:
Evaluation of the safety and antiviral activity of 3 dose levels of ACH-126,443 versus lamivudine and placebo over 12 weeks of treatment in the population is described.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B virus (HBV) infection, known to be hepatitis B surface antigen positive ≥ 6 months.
* Plasma HBV deoxyribonucleic acid level ≥ 100,000 copies/milliliter.
* Hepatitis B e-antigen positive.
* Human immunodeficiency virus negative.
* Basic hematologic and chemistry parameters within acceptable limits (defined in protocol).
* No need for excluded medications.
* Participants of reproductive capability must have utilized 2 approved forms of birth control, one of which must have been barrier protection.

Exclusion Criteria:

* Human immunodeficiency virus infection.
* Hepatitis C co-infection.
* Concurrent systemic antiviral treatment.
* Previous antiviral treatment for HBV infection within 6 months prior to randomization or treatment with lamivudine for more than 6 months at any time in the past.
* Previous therapy with agents with significant systemic myelosuppressive or cytotoxic potential within 3 months of study start or the expected need for such therapy at study start.
* Alcohol abuse.
* Pregnancy or breast-feeding.
* Inability to tolerate oral medication.
* Aspartate aminotransferase > 7.0 times the upper limit of normal.
* Alanine aminotransferase > 7.0 times the upper limit of normal.
* Any clinical condition or prior therapy that, in the Investigators opinion, would make the participant unsuitable for the study or unable to comply with the dosing requirements.
* Use of any investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2002-02; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Clinical Trial Site, Sofia, Bulgaria
- Federal Republic of Yugoslavia (2):
  - Clinical Trial Site, Belgrade
  - Clinical Trial Site, Novi Sad